CLINICAL TRIAL: NCT01651221
Title: Repeated Food Exposure Via the Olfactory and Gustatory Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 8879B
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Habituation
Keywords: gustatory response; olfactory response
MeSH Terms: conditions — Substance-Related Disorders | interventions — Habituation, Psychophysiologic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Olfactory (Experimental): Habituation of olfactory response
  Interventions: Other: Habituation
- gustatory (Experimental): Habituation of gustatory response.
  Interventions: Other: Habituation
- olfactory and gustatory (Experimental): Habituation of olfactory and gustatory response
  Interventions: Other: Habituation

INTERVENTIONS:
Other: Habituation — Habituation will be measured for each the conditions (olfactory, gustatory, olfactory and gustatory) of the study.

SUMMARY:
Increasing exposure to a single orosensory cue without ingestion of additional energy may promote an increased rate of habituation, more rapid satiation, and reduced intake. This exposure can occur via smell (olfactory) and taste (gustatory) systems.It is not clear if repeated exposure via the combined olfactory and gustatory systems increases the rate of habituation more so than repeated exposure through one of these systems. Thus, the purpose of this investigation is to examine the amount of salivation occurring in 12 trials of exposure to a food via the olfactory, gustatory, and combined olfactory and gustatory systems. The primary dependent variable will be the amount of salivation in the 12 trials. It is hypothesized that a more rapid decrease in salivation will occur across trials in the combined olfactory and gustatory exposure as compared to the other two conditions, indicating a more rapid rate of habituation.

DETAILED DESCRIPTION:
Approximately two of every three adults in the U.S. are overweight or obese. The high prevalence of overweight/obesity negatively affects the health of the population, as obese individuals are at increased risk for developing several chronic diseases.

Successful control of body weight depends on effectively regulating eating. Satiation, the process by which an eating bout ends, assists with eating regulation, and factors that quicken the onset of satiation may aid with decreasing intake. One factor believed to influence satiation is the rate of decrease in consummatory response (habituation) to repeated presentations of food orosensory cues. Habituation is a basic form of learning, in which behavioral and physiological responses decrease in response to repeated presentations of a stimulus, with the decrease in response unrelated to sensory adaptation/fatigue or motor fatigue.

In one condition, participants will smell lemon and lime across 12 trials (olfactory exposure), in another condition participants will taste the juices across 12 trials (gustatory exposure), and in the last condition participants will smell and taste the juices across 12 trials (olfactory + gustatory exposure). The primary dependent variable will be the amount of salivation in the 12 trials. It is hypothesized that a more rapid decrease in salivation will occur across trials in the combined olfactory and gustatory exposure as compared to the other two conditions, indicating a more rapid rate of habituation

ELIGIBILITY:
Inclusion Criteria:

* Dietary restraint scores of less than or equal to 12 on the Three Factor -
* Eating Questionnaire-Cognitive Restraint scale.
* Have a body mass index (BMI) between 18.5 and 24.9.

Exclusion Criteria:

* Are taking medications or having an illness which might influence salivation, smell, and taste (i.e. upper respiratory illness, methylphenidate, atropine, Benadryl, Elavil, etc)
* Are currently dieting
* Are a binge eater
* Do not at least moderately like lemon or lime flavor scoring < 50 on a 100 mm visual analogue scale
* Are a regular smoker
* Have any dietary restrictions that will inhibit participation including food allergies

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Amount of Salivation | 12 trials (90 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, PhD RD LDN, Principal Investigator — University of Tennessee
Locations (1):
- Healthy Eating and Activity Lab, University of Tennessee, Knoxville, Tennessee, United States